CLINICAL TRIAL: NCT00440752
Title: The Impact of Artemether-Lumefantrine on Genes Associated With Antimalarial Resistance in an Area of Seasonal Transmission
Brief Title: The Impact of Artemether-Lumefantrine on Genes Associated With Antimalarial Resistance
Status: Completed | Type: Observational
Sponsor: Tropical Medicine Research Institute (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); World Health Organization (Other); International Atomic Energy Agency (Other Government)
Other Study IDs: AL Oct-Dec/06-07
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2007-10

CONDITIONS: Falciparum Malaria; Antimalarials
Keywords: Artemether-lumefantrine; Plasmodium falciparum; drug resistance genes
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood spots on glass fibre membranes. 0.5ml of whole blood preserved in TRI reagent.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AL: Cohort of study participants receiving treatment with artemether-lumefantrine

SUMMARY:
The newly introduced antimalarial drug artemether-lumefantrine is currently recommended as second line antimalarial in Sudan. Recurrent infection after treatment with this drug has been associated with selection of certain genes in the malaria parasite. However there is no information on this association in Sudan.This study is going to look into the genetics of resistance to artemether-lumefantrine.

DETAILED DESCRIPTION:
In Sudan the current treatment protocol includes two artemisinin combinations (ACT); artesunate + sulphadoxine/pyrimethamine (AS/SP) as first line and artemether-lumefantrine (AL) as second line. This protocol has been implemented in 2004, since then various studies have reported the high efficacy of both combinations (e.g. Adam et al., 2005; Elamin et al., 2005; Mohamed et al., 2006).

However, there has been no report of the impact of these combinations on drug resistance markers in Sudan. Data from other African countries has shown that AL selects for certain alleles in the pfmdr-1 gene (Sisowath et al., 2005, Dokomajilar et al., 2006; Humphreys et al., 2007), but the impact on the prevalence of different pfcrt and pfmdr-1alleles remains unclear. It is essential to monitor ACT efficacy in addition to identify molecular markers that are associated with response to different drugs to facilitate epidemiological surveys for evidence based decision making. Recent work in The Gambia suggests that transmission-related endpoints, such as emergence of gametocytes after treatment, may be better indicators of emerging drug resistance (Hallett et al., 2006).

The aim of the proposed study is to examine the impact of treatment with artemether-lumefantrine (AL) on alleles of pfcrt and pfmdr-1 in P. falciparum isolates in an area of marked seasonal transmission in eastern Sudan. Most studies of resistance markers measure marker prevalence by DNA amplification, but we will also investigate gene expression using quantitative amplification of mRNA encoding pfcrt and pfmdr-1. The impact of genotype and gene expression levels on treatment outcome, and on the emergence and density of peripheral gametocytes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Mono-infection with P. falciparum by microscopy.
* Initial parasite density of 1000 to 100,000 asexual parasites/µl.
* Absence of general danger signs or other signs of severe and complicated falciparum malaria according to WHO definitions.
* Informed consent provided by patient or parent/guardian.

Exclusion Criteria:

* Pregnancy
* Infection with mixed Plasmodium sp.
* Signs of severe malaria or any danger signs
* Refusal to provide consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Levels of expression of pfcrt and pfmdr-1 alleles on day 0, 3, 7, 14, 21, 28 detected by real-time PCR. | 2007 to 2009

SECONDARY OUTCOMES:
Parasitological failure occurring at day 3, 7, 14, 21, 28 or any other day during this period. | within 28 days of subject recruitment
Gametocyte development detected by reverse transcriptase PCR on day 0, 3, 14 and 28 | 2008 to 2009

CONTACTS AND LOCATIONS:
Overall Officials: Colin Sutherland, PhD., Principal Investigator — London School of Hygiene and Tropical Medicine; Badria B El-Sayed, PhD, Study Chair — Tropical Medicine Research Institute
Locations (1):
- Tropical Medicine Research Institute, Khartoum, Khartoum State, Sudan

REFERENCES:
- [Background] Dokomajilar C, Nsobya SL, Greenhouse B, Rosenthal PJ, Dorsey G. Selection of Plasmodium falciparum pfmdr1 alleles following therapy with artemether-lumefantrine in an area of Uganda where malaria is highly endemic. Antimicrob Agents Chemother. 2006 May;50(5):1893-5. doi: 10.1128/AAC.50.5.1893-1895.2006. PMID 16641472
- [Background] Humphreys GS, Merinopoulos I, Ahmed J, Whitty CJ, Mutabingwa TK, Sutherland CJ, Hallett RL. Amodiaquine and artemether-lumefantrine select distinct alleles of the Plasmodium falciparum mdr1 gene in Tanzanian children treated for uncomplicated malaria. Antimicrob Agents Chemother. 2007 Mar;51(3):991-7. doi: 10.1128/AAC.00875-06. Epub 2006 Dec 28. PMID 17194834
- [Background] Sisowath C, Stromberg J, Martensson A, Msellem M, Obondo C, Bjorkman A, Gil JP. In vivo selection of Plasmodium falciparum pfmdr1 86N coding alleles by artemether-lumefantrine (Coartem). J Infect Dis. 2005 Mar 15;191(6):1014-7. doi: 10.1086/427997. Epub 2005 Feb 8. PMID 15717281